CLINICAL TRIAL: NCT06599346
Title: Study on the Effects of Mesenchymal Stem Cell Culture Supernatant on the Prevention and Treatment of Mucosal Injury in Hematology Patients
Brief Title: Effects of Mesenchymal Stem Cell Supernatant on Prevention and Treatment of Skin/Mucosal Injury in Hematology Patients
Acronym: MSC-MucInj
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The General Hospital of Western Theater Command (Other)
Responsible Party: Principal Investigator, Chendan, Associate Professor, The General Hospital of Western Theater Command
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023EC4-ky008
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mucositis; Hematopoietic Stem Cell Transplantation; Chemotherapy-Induced Mucositis; Radiation-Induced Mucositis
Keywords: Mesenchymal Stem Cell Supernatant; Mesenchymal Stem Cell Exosomes; Mucosal Injury; Hematopoietic Stem Cell Transplantation; Chemotherapy; Radiotherapy; Oral Mucosal Injury; Skin Mucosal Injury; Bladder Injury; HSCT Complications; Tissue Regeneration; Mucosal Repair
MeSH Terms: conditions — Mucositis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants in this study will be randomly assigned to one of two groups in parallel. The control group will receive standard care for mucosal injuries (such as oral rinses and supportive care), while the intervention group will receive MSC supernatant treatment in addition to standard care. The treatments will be administered concurrently, and both groups will be monitored for the duration of the study to assess the effectiveness and safety of MSC supernatant in healing mucosal injuries caused by HSCT, chemotherapy, and radiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Standard Care for Mucositis (Active Comparator): Participants in this arm will receive standard care for mucositis, which may include oral rinses, topical treatments, and supportive care. Standard care will be tailored based on the type and severity of the mucosal injury (oral, skin, or bladder).
  Interventions: Other: Standard Care
- Experimental: MSC Supernatant + Standard Care for Mucositis (Experimental): Participants in this arm will receive MSC supernatant in addition to standard care for mucositis. The MSC supernatant will be administered as follows:
  15 mL for oral mucosal injuries (mouthwash) Topical application for skin mucosal injuries (based on body surface area) 50 mL for bladder injuries (bladder irrigation)
  Interventions: Biological: MSC Supernatant + Standard Care

INTERVENTIONS:
Other: Standard Care — Participants in this arm will receive standard care for mucosal injuries, which may include oral rinses, topical treatments, and supportive care based on the type of injury.
  Arms: Active Comparator: Standard Care for Mucositis
Biological: MSC Supernatant + Standard Care — Participants in this arm will receive MSC supernatant in addition to standard care. MSC supernatant will be administered as follows:
  15 mL for oral mucosal injuries (mouthwash) Topical application for skin mucosal injuries (based on body surface area) 50 mL for bladder injuries (bladder irrigation)
  Arms: Experimental: MSC Supernatant + Standard Care for Mucositis

SUMMARY:
This clinical trial is studying the effects of mesenchymal stem cell (MSC) culture supernatant on the prevention and treatment of mucosal injuries in patients undergoing hematopoietic stem cell transplantation (HSCT). HSCT is a common treatment for blood-related cancers and other serious blood disorders. However, many patients experience severe damage to their mucous membranes, including the lining of the mouth, skin, and bladder, due to the high-dose chemotherapy used in the treatment process. These mucosal injuries can cause pain, increase the risk of infection, and lower the patient's quality of life.

The purpose of this study is to determine whether MSC culture supernatant can help repair mucosal injuries and improve recovery for these patients. MSC culture supernatant contains substances produced by mesenchymal stem cells that may promote healing and reduce inflammation. These substances could potentially repair tissue without the risks associated with using live cells.

Participants in this trial will be randomly assigned to one of two groups: one group will receive standard care, and the other will receive MSC culture supernatant as part of their treatment. The study will look at how well MSC supernatant helps heal mucosal injuries, as well as its safety and any side effects that may occur. The outcomes of this study could lead to new ways to prevent and treat mucosal injuries in patients undergoing HSCT, improving their quality of life during and after treatment.

The trial will include 120 patients who have undergone HSCT and experienced mucosal injuries. The study will last approximately five years, from October 2020 to September 2025. Participants will be monitored throughout the trial for safety and effectiveness of the treatment, with follow-up visits scheduled to assess their progress.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the efficacy and safety of mesenchymal stem cell (MSC) culture supernatant in the prevention and treatment of mucosal injuries in patients undergoing hematopoietic stem cell transplantation (HSCT). HSCT is a critical therapy for blood-related cancers and severe hematological disorders but is often associated with significant mucosal injuries caused by the high-dose chemotherapy and radiation therapy used during the preconditioning phase. These injuries predominantly affect the oral mucosa, skin, and bladder, resulting in severe pain, elevated infection risks, and prolonged hospitalization.

Current treatment options for mucosal injuries focus on symptom management but provide limited efficacy in accelerating tissue repair or preventing further complications. MSC culture supernatant contains a variety of bioactive factors, including growth factors and cytokines secreted by MSCs during culture. These factors are believed to promote tissue repair and regeneration, offering a promising alternative to live cell therapies, which pose higher safety risks. This study investigates MSC supernatant as a novel therapeutic option for mucosal injuries in HSCT patients.

Study Design:

This is a prospective, randomized controlled trial with a target enrollment of 120 patients. Participants will be randomly assigned to one of two groups:

Control Group: Patients will receive standard care for mucosal injuries, which may include oral rinses, pain management, and supportive care.

Intervention Group: Patients will receive MSC culture supernatant in addition to standard care. The MSC supernatant will be administered based on the type of mucosal injury:

Oral Mucosal Injuries: 15 mL of MSC supernatant will be used as a mouthwash. Skin Mucosal Injuries: MSC supernatant will be applied topically, proportional to the affected body surface area.

Bladder Injuries (Cystitis): 50 mL of MSC supernatant will be used for bladder irrigation.

Study Objectives:

Primary Objective: To assess the efficacy of MSC culture supernatant in the healing of mucosal injuries in HSCT patients. Mucosal healing will be evaluated using standardized scales such as the WHO mucosal injury scale and patient-reported pain scores.

Secondary Objective: To determine the safety and tolerability of MSC supernatant by monitoring adverse events (AEs) and serious adverse events (SAEs) in accordance with the CTCAE v5.0 criteria.

Exploratory Objectives: To explore the impact of MSC supernatant on tissue repair, infection reduction, length of hospital stay, and patient quality of life (QoL) during recovery from HSCT.

Inclusion and Exclusion Criteria:

Inclusion Criteria:

Patients who have undergone HSCT and developed mucosal injuries (oral, skin, or bladder).

Ability to understand and provide informed consent, and comply with study requirements.

Exclusion Criteria:

Patients with severe organ dysfunction or uncontrolled active infections. Patients with known allergies to MSC supernatant. Pregnant or breastfeeding women. Patients who are HIV-positive or have active hepatitis B or C. Patients enrolled in another clinical trial within the last four weeks.

Outcome Measures:

Primary Outcome: Mucosal injury healing, defined as a reduction in the mucosal injury grade to ≤1 and a pain score of ≤2.

Secondary Outcomes: Frequency and severity of adverse events related to MSC supernatant, measured according to CTCAE v5.0.

Exploratory Outcomes: Reduction in infection rates, shortened hospital stays, and improved patient-reported quality of life (QoL).

Monitoring and Safety:

Participants will undergo regular evaluations, including weekly assessments during the treatment phase and monthly follow-ups post-treatment. Laboratory tests (e.g., blood counts, liver and kidney function tests) and vital signs will be closely monitored to ensure patient safety. Adverse events will be documented, and appropriate interventions will be implemented as required.

It is important to note that while no Data Monitoring Committee (DMC) has been established for this study, safety oversight will be conducted by the research team following standard safety monitoring protocols.

Study Duration:

The trial is set to run from October 2020 to September 2025, with data collection for the primary outcomes expected to be completed by September 2025. Participants will be followed for the entirety of the study period, and long-term assessments will be conducted to evaluate the sustained efficacy and safety of MSC supernatant for mucosal injuries.

Significance:

This trial has the potential to introduce an innovative treatment strategy for managing mucosal injuries in HSCT patients. By utilizing the bioactive components of MSC culture supernatant, this therapy may enhance tissue regeneration, lower infection risk, and expedite recovery. If proven effective, this treatment could significantly improve patient outcomes and overall quality of life during and after HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older.
* Patients who have undergone hematopoietic stem cell transplantation (HSCT).
* Patients who have developed mucosal injuries (oral, skin, or bladder) after HSCT, chemotherapy, or radiotherapy.
* Patients who are willing to provide informed consent and comply with the study procedures.

Exclusion Criteria:

* Patients with severe organ dysfunction (e.g., heart, liver, kidney failure) that could interfere with the study.
* Patients with uncontrolled active infections.
* Known allergies or hypersensitivity to MSC supernatant.
* Pregnant or breastfeeding women.
* Patients with HIV or active hepatitis B or C infections.
* Patients who have participated in another clinical trial within the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Mucosal Injury Healing | 8 weeks after the start of treatment.
  The degree of mucosal injury healing will be assessed using the WHO Mucosal Injury Scale (World Health Organization Mucosal Injury Grading Scale) and a pain score measured by the Visual Analog Scale (VAS) for pain.
  WHO Mucosal Injury Scale: This scale assesses mucosal injury severity. The grades range from 0 (no injury) to 4 (severe ulceration and bleeding). A lower score indicates better mucosal health.
  Visual Analog Scale (VAS) for pain: This scale measures pain on a range of 0 (no pain) to 10 (worst pain imaginable). A lower score indicates less pain.
  The outcome will measure the percentage of participants with WHO mucosal injury grades ≤1 and VAS pain scores ≤2, indicating mild or no injury and low pain.

SECONDARY OUTCOMES:
Mucosal Infection Rates | From the start of treatment through 8 weeks post-treatment.
  The number of participants developing secondary infections related to mucosal injuries (oral, skin, bladder) during the study period. This outcome will report infection rates as a percentage of participants.
Hospital Stay Duration | From the start of treatment until discharge, assessed up to 12 weeks.
  The number of days participants remain hospitalized during the study will be tracked, with comparisons made between the control and intervention groups.

OTHER OUTCOMES:
Patient Quality of Life (QoL) | 12 weeks after the start of treatment.
  Assessed using the EQ-5D Questionnaire (5 dimensions, scores range from 5 to 25). Lower scores indicate better quality of life.
  Participants will also rate overall health using the VAS, ranging from 0 (worst) to 100 (best). Higher scores indicate better health.
  Additionally, participants will rate their overall health using a Visual Analog Scale (VAS), ranging from 0 (worst imaginable health) to 100 (best imaginable health), where higher scores indicate better health.
  Scale: The EQ-5D uses a scale from 1 (no problems) to 5 (extreme problems) for each of the five dimensions. The total score ranges from 5 to 25, with lower scores indicating a better quality of life.
  Participants will also rate overall health using the VAS, ranging from 0 (worst) to 100 (best). Higher scores indicate better health.
  EQ-5D: The scale ranges from 1 (no problems) to 5 (extreme problems) across each dimension, with a total score ranging from 5 to 25. Lower scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Chen, Bachelor, Principal Investigator — Department of Hematology, The General Hospital of Western Theater Command; Hao Yao, Ph.D, Principal Investigator — Department of Hematology, The General Hospital of Western Theater Command
Locations (1):
- Department of Hematology, The General Hospital of Western Theater Command, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No